CLINICAL TRIAL: NCT05400889
Title: Real-world Experience With Inhibitors of Janus Kinase for the Treatment of Idiopathic Inflammatory Myopathies -- a Prospective Observational Study
Brief Title: Clinical Characteristics and Mechanism Research of Inhibitors of Janus Kinase in the Idiopathic Inflammatory Myopathies
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, HeJing, Professor, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20220420 JAKi-IIM
Record Dates: First submitted 2022-05-16; First posted 2022-06-02 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Idiopathic Inflammatory Myopathies
MeSH Terms: conditions — Myositis | interventions — tofacitinib; baricitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- tofacitinib or baricitinib (Experimental): Tofacitinib 5mg was taken orally once or twice a day and baricitinib 2mg or 4mg was taken orally once a day for 6 months.
  Interventions: Drug: tofacitinib

INTERVENTIONS:
Drug: tofacitinib — Tofacitinib 5mg was taken orally once or twice a day and baricitinib 2mg or 4mg was taken orally once a day for 6 months.
  Other Names: Baricitinib

SUMMARY:
This study aims to explore the clinical characteristics and mechanism of inhibitors of janus kinase in the treatment of idiopathic inflammatory myopathies

DETAILED DESCRIPTION:
The investigators designed a single center, open-label, prospective study. Adults with active idiopathic inflammatory myopathies will be enrolled, meeting the Bohan & Peter Dermatomyositis/Polymyositis(DM/PM) or Rheumatology(ACR) & European allance of associations for rheumatology(EULAR)(2017) diagnostic criteria. Inhibitors of janus kinase including tofacitinib 5 mg once a day or twice a day and baricitinib 2mg once a day or 4mg once a day was administered for 6 months to explore its efficacy and safety, which could help to evaluate inhibitors of janus kinase's clinical characteristics and mechanism. Patients would be evaluated the improvement of clinical and laboratory indexes. Changes of symptoms, immune cell subsets and cytokines were monitored. Symptoms were evaluated by Visual Analogue Scale (VAS) of patient global and physician global, manual muscle testing(MMT-8), the Health Assessment Questionnaire(HAQ), Creatine kinase, Myositis Disease Activity Assessment Tool(MDAAT).

ELIGIBILITY:
Inclusion Criteria:

* Adults between 18 years and 75 years of age.
* Adults with active idiopathic inflammatory myopathies will be enrolled, meeting the Bohan & Peter DM/PM or American College of Rheumatology(ACR) & European allance of associations for rheumatology(EULAR)(2017) diagnostic criteria.
* Written informed consent should be obtained from each study subject.
* Concomitant immunosuppressive agents or glucocorticoids were allowed, but subjects should have been on these therapies at least 4 weeks and on a stable dose for ≥4 weeks(glucocorticoid doses are lower than <0.5mg/kg/d).
* Consent to use effective contraception during the study (women of childbearing age).

Exclusion Criteria:

Any subject meeting either of the following criteria should be excluded:

* Laboratory abnormality: Hb<8 g/dl or platelet<60*10^9/L, or combined with severe hepatic, renal and cardiac insufficiency;
* Myositis in overlap with another systemic autoimmune rheumatic disorder, cancer-associated myositis, inclusion body myositis or any other non-immune mediated myopathy.
* Biologics such as rituximab are not allowed in the 3-month before enrollment.
* Patients with malignancy within 3 years of screening.
* Patients with hypersensitivity to study drug.
* Active infections(including but not limited to hepatitis, HIV).
* Uncontrolled mental or emotional disorders.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-06-10 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Immunological Responses | week 24
  Changes of follicular helper T cells (TFH) before and after tofacitinib treatment are analysed to evaluate efficacy.

SECONDARY OUTCOMES:
Myositis Disease Activity Assessment Tool(MDAAT) | week 24
  Change of MDAAT(Myositis Disease Activity Assessment Tool) is measurement of effectiveness. MDAAT ranges from 0 to 10cm. The more severe the disease activity, the higher the score. We define response as an improvement of MDAAT at least 5%.

CONTACTS AND LOCATIONS:
Overall Officials: Zhanguo Li, Principal Investigator — Peking University Institute of Rheuamotology and Immunology
Locations (1):
- Department of Rheumatology and Immunology, Peking University People's Hospital, Beijing, Beijing Municipality, China